CLINICAL TRIAL: NCT01315743
Title: Team COOL Pilot Study
Acronym: Team COOL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0601S79069
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Multicomponent School Based Behavioral Intervention; Prevent Further Weight Gain and or Promote; Weight Loss Among Adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Team COOL

INTERVENTIONS:
Behavioral: Team COOL — 1) a classroom-based experiential curriculum that incorporated school, family and community-linked activities to promote physical activity, healthy eating and limited television viewing, 2) environmental modifications of food and beverage offerings and physical activity opportunities at school and 3) a teacher-guided, youth-directed health advisory council to promote and support physical activity, healthy eating and limited television viewing.

SUMMARY:
The goal of this exploratory pilot study was to develop and test the acceptability and feasibility of an innovative alternative high school-based intervention to prevent further weight gain and/or promote weight loss among a sample of ethnically and economically diverse adolescents.

DETAILED DESCRIPTION:
The goal of this exploratory pilot study was to develop and test the acceptability and feasibility of an innovative alternative high school-based intervention to prevent further weight gain and/or promote weight loss among a sample of ethnically and economically diverse adolescents. The proposed study will use a group randomized trial design and target boys and girls, ages 15-20 years old, attending six alternative high schools in the Minneapolis-St Paul metropolitan area. Alternative high schools are public or private schools that offer a nontraditional educational experience for at-risk students, such as dropouts, expelled students, truants and hard to reach learners who have not succeeded in regular school systems. Although low levels of physical activity (PA) and unhealthy dietary practices, behaviors regarded as a primary cause of the overweight/obesity epidemic among youth, are prevalent among teens attending alternative schools, school-based programs targeting these behaviors have not been tested and evaluated.

Three schools were randomized to the intervention/treatment condition and three schools to a minimal intervention/comparison condition. Social Cognitive Theory and ecological theory provided the theoretical basis for the multi-component intervention, which included 1) a classroom-based experiential curriculum that incorporated school, family and community-linked activities to promote physical activity, healthy eating and limited television viewing, 2) environmental modifications of food and beverage offerings and physical activity opportunities at school and 3) a teacher-guided, youth-directed health advisory council to promote and support physical activity, healthy eating and limited television viewing.

Student and school-level measurements were taken at baseline, 6 months post randomization and at the completion of the 18 month intervention. Student-level measures included a self-administered psychosocial survey, the 3-day Previous Day Physical Activity Report and moderate-to-vigorous physical activity levels of students as measured by an Actigraph accelerometer. School-level measures assessed the availability of physical activity opportunities and healthy foods at school.

Hypothesis: Adolescents attending alternative high schools will report high participation rates and a high degree of satisfaction with a multi-component school-based intervention targeting students' PA, diet and TV viewing practices.

ELIGIBILITY:
Inclusion Criteria:

Because this research is a group randomized trial, eligibility criteria were based primarily on school characteristics rather than student characteristics. Schools eligible for recruitment were required to: 1) identify as either an area learning center (ALC), alternative learning program (ALP) or contracted alternative, 2) be open year around (a requirement for all state ALCs; an option for ALPs), 3) enroll 11th and 12th grade students, 4) project a September 2006 enrollment of 75 students, 5) require student attendance on campus at least 10 hours/week and 6) have access to an indoor facility for physical activity. Therefore, all students attending a participating school were eligible to take part in the study and exclusion will occur only in case of parental or student denial of consent. Students and parents/guardians of students who were not fluent in English were not included in measurement.

-

Exclusion Criteria: Alternative programs that serve primarily pregnant and disabled teens or function exclusively as day treatment programs for juvenile offenders were not eligible to participate in this study.Students and parents/guardians of students who were not fluent in English were not included in measurement.

-

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

REFERENCES:
- [Derived] Arcan C, Kubik MY, Fulkerson JA, Hannan PJ, Story M. Substance use and dietary practices among students attending alternative high schools: results from a pilot study. BMC Public Health. 2011 Apr 25;11:263. doi: 10.1186/1471-2458-11-263. PMID 21518437